CLINICAL TRIAL: NCT01204853
Title: A Phase 3, Multi-Center, Open Label Study To Evaluate The Safety And Efficacy Of Sitaxentan Sodium In Japanese Subjects With Pulmonary Arterial Hypertension
Brief Title: A 12 Week Safety And Efficacy Study Of Sitaxentan Sodium In Japanese Pulmonary Arterial Hypertension Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Safety Issue: The trial was prematurely terminated on Dec 9, 2010, due to safety concerns, specifically new emerging evidence of hepatic injury.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1321052
Record Dates: First submitted 2010-08-06; First posted 2010-09-17 (Estimated); Results first posted 2011-12-01 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-10

CONDITIONS: Hypertension, Pulmonary
Keywords: sitaxentan sodium hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — sitaxsentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sitaxentan treatment (Experimental)
  Interventions: Drug: Sitaxentan

INTERVENTIONS:
Drug: Sitaxentan — sitaxentan sodium 100 mg

SUMMARY:
The safety and efficacy at 100 mg once daily for oral dose of sitaxentan sodium were demonstrated in the STRIDE clinical trial program. Sitaxentan sodium was approved in the EU, Canada and Australia. In this study, the safety and efficacy after administrations of sitaxentan sodium at a dose of 100 mg alone or in combination with another medication will be investigated in Japanese PAH patients.

ELIGIBILITY:
Inclusion Criteria:

* Has a current diagnosis of symptomatic PAH
* Has 6MWT distances from 150 to 450 meters and distance

Exclusion Criteria:

* Previous exposure to an endothelin receptor antagonist
* Has uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure >160 mm Hg or sitting diastolic blood pressure >100 mm Hg at Screening.
* Has hypotension defined as systolic arterial pressure <90 mm Hg after sitting for 5 minutes at Screening.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Japan (2):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Shinjyuku-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321052&StudyName=A%2012%20Week%20Safety%20And%20Efficacy%20Study%20Of%20Sitaxentan%20Sodium%20In%20Japanese%20Pulmonary%20Arterial%20Hypertension%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitaxentan Treatment: All participants received one 100 mg film-coated tablet of sitaxentan daily for 12 weeks. Participants who had already received a stable dose of pulmonary arterial hypertension (PAH)-specific drug (sildenafil or beraprost) for at least 3 month prior to screening, continued to receive the PAH-specific drug during study period.
Period: Overall Study
Arm/Group | Sitaxentan Treatment
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 2
Age, Customized [Number; unit: Participant]
  <=18 years | 0
  19-64 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with any adverse events, severe adverse events, serious adverse events
Time Frame: 12 weeks
Population: Safety analysis set is defined as all participants who receive at least one dose of the study drug.
  Descriptive statistics for adverse events were not calculated due to a small number of subjects.
Measure: Number; unit: Participant
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 2
Participant
  All-causality adverse events | 1
  All-causality serious adverse events | 0
  All-causality severe adverse events | 0

2. Primary Outcome: Change From Baseline in 6-minute Walk Distance
Description: Change from baseline in 6-minute walk distance is calculated as the value at Week 12 minus value at baseline.
Time Frame: 12 weeks
Population: Efficacy analysis set is defined as all participants who receive at least one dose of the study drug and had efficacy observations at baseline in any efficacy assessments.
  Descriptive statistics for change from baseline in 6-minute walk distance were not calculated due to a small number of participants.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in WHO Functional Class
Description: The change from baseline in WHO functional class was classified into "Improved", "No change" and "Worsened". The change from baseline in WHO functional class at Week 12 was to be summarized with frequency count and percentage in each category based on imputed data for missing values at Week 12.
Time Frame: 12 weeks
Population: Efficacy analysis set is defined as all participants who receive at least one dose of the study drug and had efficacy observations at baseline in any efficacy assessments.
  Descriptive statistics for change from baseline in WHO functional class were not calculated due to a small number of participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Haemodynamics Parameters
Description: The following haemodynamic measurements were assessed: right arterial pressure, pulmonary arterial systolic pressure, pulmonary arterial diastolic pressure, mean pulmonary arterial pressure, pulmonary capillary wedge pressure, left ventricular-end diastolic pressure, cardiac output, systemic arterial blood pressure (systolic, diastolic and mean), and heart rate.
  Change from baseline in haemodynamics parameters is calculated as the value at Week 12 minus value at baseline.
Time Frame: 12 weeks
Population: Efficacy analysis set is defined as all participants who receive at least one dose of the study drug and had efficacy observations at baseline in any efficacy assessments.
  Descriptive statistics for change from baseline in haemodynamics parameters were not calculated due to a small number of participants.
Measure: Number; unit: Participants
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in N-amino Terminal Fragment of the Prohormone Brain Natriuretic Peptide (NT-pro BNP)
Description: Change from baseline in NT-pro BNP is calculated as the value at Week 12 minus value at baseline.
Time Frame: 12 weeks
Population: Efficacy analysis set is defined as all participants who receive at least one dose of the study drug and had efficacy observations at baseline in any efficacy assessments.
  Descriptive statistics for change from baseline in NT-pro BNP were not calculated due to a small number of participants.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Clinical Worsening
Description: Clinical worsening is defined as 1) Hospitalization for worsening pulmonary arterial hypertension, 2) On-study death, 3) Heart-lung or lung transplantation, 4) Atrial septostomy, 5) Addition of the chronic medications for the treatment of worsening pulmonary arterial hypertension, and 6) Initiation of oxygen.
Time Frame: 12 weeks
Population: Efficacy analysis set is defined as all participants who receive at least one dose of the study drug and had efficacy observations at baseline in any efficacy assessments.
  Descriptive statistics for clinical worsening were not calculated due to a small number of participants.
Measure: Number; unit: Participants
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Pharmacokinetic (PK) Parameters at Steady State
Description: The following PK parameters at the steady state were evaluated: maximum observed concentration during the dosing interval (Cmax), time for maximum observed concentration during the dosing interval (Tmax), area under the plasma concentration-time curve over dosing interval tau for multiple dose (AUCtau), terminal elimination half-life (t1/2), apparent clearance (CL/F) and apparent volume of distribution during the terminal elimination phase (Vz/F) at Week 12/Termination (as data permit), and concentration predose during multiple dosing (Ctrough) at Week 2, 4, 8 and 12/Termination.
Time Frame: pre-dose at Week 2, 4, 8, and pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24 hours post-dose at Week 12 or study termination
Population: The PK concentration set was defined as all participants who have at least 1 concentration.
  The PK parameter analysis set was defined as all participants who have at least 1 of PK parameters of interest.
  Descriptive statistics for PK parameters were not calculated due to a small number of participants.
Measure: Number; unit: Participants
Arm/Group | Sitaxentan Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sitaxentan Treatment
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxentan Treatment (N=2)
Abdominal pain (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Oedema (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Panic attack (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.